CLINICAL TRIAL: NCT01957579
Title: A Phase 1, Dose-escalation Study of MEDI-551, a Humanized Monoclonal Antibody Directed Against CD19, in Japanese Adult Patients With Relapsed or Refractory Advanced B-cell Malignancies
Brief Title: A Phase 1, Dose-escalation Study of MEDI-551 in Japanese Adult Patients With Relapsed or Refractory Advanced B-cell Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D2850C00001; NCT01377116 (obsolete NCT alias)
Record Dates: First submitted 2013-10-01; First posted 2013-10-08 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2017-06-12 (Actual); Status verified 2017-05

CONDITIONS: Blood Cancer; Advanced B Cell Malignancies
Keywords: Phase I; advanced; B cell malignancies; dose escalation; CD19; Japanese
MeSH Terms: conditions — Hematologic Neoplasms | interventions — inebilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MEDI-551 (Experimental)
  Interventions: Drug: MEDI-551

INTERVENTIONS:
Drug: MEDI-551 — MEDI-551 will be administered by intravenous infusion at dose of 2, 4 or 8 mg/kg once per week on Days 1 and 8 in the first cycle and then once every 28 days at the start of each subsequent cycle

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of MEDI-551 in Japanese patients with relapsed or refractory advanced B-cell malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Japanese men or women at least 20 years of age
* Histologically confirmed CLL (excluding small lymphocytic lymphoma (SLL)), DLBCL, FL, or MM.
* Karnofsky Performance Status ≥70;
* Life expectancy of ≥12 weeks

Exclusion Criteria:

* Any available standard line of therapy known to be life-prolonging or life-saving
* Any concurrent chemotherapy, radiotherapy, immunotherapy, biologic or hormonal therapy for treatment of cancer
* Previous therapy directed against CD19, such as monoclonal antibodies or MAb conjugates

Ages: 20 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-05-25 (Actual); Primary Completion 2015-09-15 (Actual); Study Completion 2015-09-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Japan (3):
  - Research Site, Fukuoka
  - Research Site, Isehara-shi
  - Research Site, Nagoya

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled on 25 May 2011. Last patient last visit on 15 September 2015.
Pre-assignment Details: A total of 32 patients were enrolled into the study. Twelve patients were screen failures, thus 20 patients received MEDI-551.
Groups:
- 2 mg/kg: MEDI-551 2 mg/kg
- 4 mg/kg: MEDI-551 4 mg/kg
- 8 mg/kg: MEDI-551 8 mg/kg
- 12 mg/kg: MEDI-551 12 mg/kg
Period: Overall Study
Arm/Group | 2 mg/kg | 4 mg/kg | 8 mg/kg | 12 mg/kg
Started | 3 | 7 | 4 | 6
Completed | 3 | 6 | 2 | 6
Not Completed | 0 | 1 | 2 | 0
Not completed — Withdrawal of concent | 0 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: All patients who received at least 1 dose of MEDI-551.
Groups:
- 2 mg/kg: MEDI-551 2mg/kg
- Total: Total of all reporting groups
Arm/Group | 2 mg/kg | 4 mg/kg | 8 mg/kg | 12 mg/kg | Total
Number analyzed (Participants) | 3 | 7 | 4 | 6 | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.3 (8.1) [43 to 59] | 57.4 (10.5) [41 to 70] | 67.0 (8.7) [54 to 72] | 67.3 (11.4) [54 to 83] | 61.3 (11.4) [41 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 0 | 3 | 10
  Male | 1 | 2 | 4 | 3 | 10
Disease Type [Number; unit: Participants] — Disease Type (CLL: chronic lymphocytic leukemia, DLBCL: diffuse large B-cell lymphoma, FL: follicular lymphoma, MM: multiple myeloma)
  Participants
    CLL | 1 | 0 | 0 | 1 | 2
    DLBCL | 0 | 2 | 2 | 2 | 6
    FL | 2 | 4 | 2 | 3 | 11
    MM | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Time Frame: From baseline to 30 days after the last dose of study drug
Population: All patients who received at least 1 dose of MEDI-551.
Measure: Number; unit: Participants
Arm/Group | 2 mg/kg | 4 mg/kg | 8 mg/kg | 12 mg/kg
Number analyzed (Participants) | 3 | 7 | 4 | 6
Participants
  At least 1 Adverse Events (AE) | 3 | 6 | 4 | 6
  At least 1 AE of CTCAE Grade 3 or higher | 2 | 2 | 1 | 3
  At least 1 Serious Adverse Events (SAE) | 1 | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With Dose Limiting Toxicities
Description: A MEDI-551 treatment-related AE of any toxicity grade that lead to an inability to receive a full cycle (2 doses) of MEDI-551, or, any Grade 3 or higher toxicity that could not be reasonably ascribed to another cause, such as disease progression or accident.
Time Frame: From baseline to 28 days after the first dose of study drug
Population: All subjects in the dose escalation phase who have received MEDI-551 at Day 1 and Day 8 and completed the safety follow-up through the dose-limiting toxicity (DLT) evaluation period (28 days), or who experienced a DLT.
Measure: Number; unit: Participants
Arm/Group | 2 mg/kg | 4 mg/kg | 8 mg/kg | 12 mg/kg
Number analyzed (Participants) | 3 | 6 | 3 | 6
Participants
  At least 1 Dose Limiting Toxicity | 0 | 1 | 0 | 2
  CTCAE Grade 3 or higher non-hematologic toxicity | 0 | 1 | 0 | 1
  CTCAE Grade 3 or higher hematologic toxicity | 0 | 0 | 0 | 1

3. Secondary Outcome: Maximum Tolerated Dose
Description: A dose was considered non-tolerated and dose escalation stopped if ≥2 of up to 6 evaluable patients experienced a DLT at any dose level. MTD is the last dose level before the non-tolerated dose.
Time Frame: From baseline to 28 days after the first dose of study drug
Population: as for outcome 2
Measure: Number; unit: mg/kg
Groups:
- MEDI-551: MEDI-551 2, 4, 8 and 12 mg/kg were evaluated
Arm/Group | MEDI-551
Number analyzed (Participants) | 18
mg/kg | 8

4. Secondary Outcome: MEDI-551 Trough Concentration Levels at Day 0 (Pre-dose)
Description: Lower limit of quantification for MEDI-551 was 0.1 μg/mL.
Time Frame: Day 0 (pre-dose)
Population: Patients who have trough concentration data at Day 0 (pre-dose)
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | 2 mg/kg | 4 mg/kg | 8 mg/kg | 12 mg/kg
Number analyzed (Participants) | 3 | 7 | 4 | 6
μg/mL | NA (NA) — Below limit of quantification | NA (NA) — Below limit of quantification | NA (NA) — Below limit of quantification | NA (NA) — Below limit of quantification

5. Secondary Outcome: MEDI-551 Trough Concentration Levels at Day 7
Description: Lower limit of quantification for MEDI-551 was 0.1 μg/mL.
Time Frame: Day 7
Population: Patients who have trough concentration data at Day 7
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | 2 mg/kg | 4 mg/kg | 8 mg/kg | 12 mg/kg
Number analyzed (Participants) | 3 | 6 | 4 | 4
μg/mL | 21.3 (8.65) | 39.2 (9.13) | 91.9 (31.1) | 104 (29.0)

6. Secondary Outcome: MEDI-551 Trough Concentration Levels at Day 28
Description: Lower limit of quantification for MEDI-551 was 0.1 μg/mL.
Time Frame: Day 28
Population: Patients who have trough concentration data at Day 28
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | 2 mg/kg | 4 mg/kg | 8 mg/kg | 12 mg/kg
Number analyzed (Participants) | 3 | 5 | 3 | 4
μg/mL | 23.2 (5.82) | 36.2 (5.34) | 103 (29.0) | 115 (21.3)

7. Secondary Outcome: MEDI-551 Trough Concentration Levels at Day 56
Description: Lower limit of quantification for MEDI-551 was 0.1 μg/mL.
Time Frame: Day 56
Population: Patients who have trough concentration data at Day 56
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | 2 mg/kg | 4 mg/kg | 8 mg/kg | 12 mg/kg
Number analyzed (Participants) | 3 | 5 | 3 | 4
μg/mL | 22.0 (4.92) | 33.2 (6.92) | 89.5 (13.9) | 114 (33.1)

8. Secondary Outcome: MEDI-551 Trough Concentration Levels at Day84
Description: Lower limit of quantification for MEDI-551 was 0.1 μg/mL.
Time Frame: Day 84
Population: Patients who have trough concentration data at Day 84
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | 2 mg/kg | 4 mg/kg | 8 mg/kg | 12 mg/kg
Number analyzed (Participants) | 3 | 4 | 3 | 4
μg/mL | 21.7 (4.40) | 33.7 (4.24) | 91.6 (9.25) | 103 (26.3)

9. Secondary Outcome: MEDI-551 Trough Concentration Levels at Day 112
Description: Lower limit of quantification for MEDI-551 was 0.1 μg/mL.
Time Frame: Day 112
Population: Patients who have trough concentration data at Day 112
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | 2 mg/kg | 4 mg/kg | 8 mg/kg | 12 mg/kg
Number analyzed (Participants) | 3 | 4 | 2 | 4
μg/mL | 22.9 (3.10) | 35.3 (5.07) | 85.5 (NA) — Standard Deviation was calculated only if n>=3. | 114 (64.4)

10. Secondary Outcome: MEDI-551 Trough Concentration Levels at Day 140
Description: Lower limit of quantification for MEDI-551 was 0.1 μg/mL.
Time Frame: Day 140
Population: Patients who have trough concentration data at Day 140
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | 2 mg/kg | 4 mg/kg | 8 mg/kg | 12 mg/kg
Number analyzed (Participants) | 2 | 4 | 2 | 4
μg/mL | 22.1 (NA) — Standard Deviation was calculated only if n>=3. | 36.3 (10.5) | 86.1 (NA) — Standard Deviation was calculated only if n>=3. | 117 (62.0)

11. Secondary Outcome: MEDI-551 Trough Concentration Levels at Day 168
Description: Lower limit of quantification for MEDI-551 was 0.1 μg/mL.
Time Frame: Day 168
Population: Patients who have trough concentration data at Day 168
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | 2 mg/kg | 4 mg/kg | 8 mg/kg | 12 mg/kg
Number analyzed (Participants) | 2 | 3 | 2 | 2
μg/mL | 20.0 (NA) — Standard Deviation was calculated only if n>=3. | 31.4 (8.30) | 94.1 (NA) — Standard Deviation was calculated only if n>=3. | 82.1 (NA) — Standard Deviation was calculated only if n>=3.

12. Secondary Outcome: Anti-MEDI-551 Antibodies
Description: Only 1 patient was tested positive for ADA at pre-dose of Cycle 1 Day 1. However, it was considered as false-positive because the titer value was close to the cut point, and this patient was tested negative for ADA at all subsequent cycles post-baseline.
Time Frame: From baseline to 30 days after the last dose of study drug
Population: Patients who have at least one post-baseline sample for Anti-MEDI-551 antibodies.
Measure: Number; unit: Participants
Arm/Group | 2 mg/kg | 4 mg/kg | 8 mg/kg | 12 mg/kg
Number analyzed (Participants) | 3 | 7 | 4 | 6
Participants
  positive at least 1 time point | 0 | 0 | 1 | 0
  negative at all time points | 3 | 7 | 3 | 6

13. Secondary Outcome: Number of Participants With Tumour Response in FL Patients
Description: Tumour response is defined as complete remission (CR) or partial remission (PR) (Cheson BD et al 2007).
  CR: Nodal Masses: (a) FDG-avid or PET positive prior to therapy; mass of any size permitted if PET negative; (b) Variably FDG-avid or PET negative; regression to normal size on CT; Spleen, Liver: Not palpable, nodules disappeared. Bone Marrow: Infiltrate cleared on repeat biopsy; if indeterminate by morphology, immunohistochemistry should be negative.
  PR: Nodal Masses: ≥50% decrease in sum of the product of the diameters (SPD) of up to 6 largest dominant masses; no increase in size of other nodes; (a) FDG-avid or PET positive prior to therapy; ≥1 PET positive at previously involved site; (b) Variably FDG-avid or PET negative; regression on CT. Spleen, Liver: ≥50% decrease in SPD of nodules (for single nodule in greatest transverse diameter); no increase in size of liver or spleen. Bone Marrow: Irrelevant if positive prior to therapy; cell type should be specified.
Time Frame: From the baseline to 30 days after the last dose of study drug
Population: All patients with FL who received at least 1 dose of MEDI-551 and completed at least 1 post-baseline disease assessment.
Measure: Number; unit: Participants
Groups:
- 2 mg/kg (FL): FL patients in MEDI-551 2 mg/kg cohort
- 4 mg/kg (FL): FL patients in MEDI-551 4 mg/kg cohort
- 8 mg/kg (FL): FL patients in MEDI-551 8 mg/kg cohort
- 12 mg/kg (FL): FL patients in MEDI-551 12 mg/kg cohort
Arm/Group | 2 mg/kg (FL) | 4 mg/kg (FL) | 8 mg/kg (FL) | 12 mg/kg (FL)
Number analyzed (Participants) | 2 | 4 | 2 | 3
Participants | 2 | 3 | 2 | 2

14. Secondary Outcome: Number of Participants With Tumour Response in DLBCL Patients
Description: as for outcome 13
Time Frame: From the baseline to 30 days after the last dose of study drug
Population: All patients with DLBCL who received at least 1 dose of MEDI-551 and completed at least 1 post-baseline disease assessment.
Measure: Number; unit: Participants
Groups:
- 2 mg/kg (DLBCL): DLBCL patients in MEDI-551 2 mg/kg cohort
- 4 mg/kg (DLBCL): DLBCL patients in MEDI-551 4 mg/kg cohort
- 8 mg/kg (DLBCL): DLBCL patients in MEDI-551 8 mg/kg cohort
- 12 mg/kg (DLBCL): DLBCL patients in MEDI-551 12 mg/kg cohort
Arm/Group | 2 mg/kg (DLBCL) | 4 mg/kg (DLBCL) | 8 mg/kg (DLBCL) | 12 mg/kg (DLBCL)
Number analyzed (Participants) | 0 | 2 | 2 | 2
Participants |  | 0 | 1 | 2

15. Secondary Outcome: Number of Participants With Tumour Response in CLL Patients
Description: Tumour response is defined as complete remission (CR) or partial remission (PR) (Hallek M et al 2008).
  CR: all of the following criteria have to be met, and patients have to lack disease-related constitutional symptoms; Lymphadenopathy: None; Hepatomegaly: None; Splenomegaly: None; Blood lymphocytes: <4000/μL; Marrow: Normocellular, <30%lymphocytes, no B-lymphoid nodules, hypocellular marrow defines CR with incomplete marrow recovery; Platelet count: >100000/μL; Hemoglobin: >11.0 g/dL; Neutrophils: >1500/μL PR: at least 2 of the criteria of group A plus 1 of the criteria of group B have to be met.
  Group A: Lymphadenopathy: Decrease ≥50%; Hepatomegaly: Decrease ≥50%; Splenomegaly: Decrease ≥50%; Blood lymphocytes: Decrease ≥50% from baseline; Marrow: 50% reduction in marrow infiltrate, or B-lymphoid nodules.
  Group B: Platelet count: 100000/μL or increase ≥50% over baseline; Hemoglobin: >11.0 g/dL or increase ≥50% over baseline; Neutrophils: >1500/μL or >50% improvement over baseline.
Time Frame: From the baseline to 30 days after the last dose of study drug
Population: All patients with CLL who received at least 1 dose of MEDI-551 and completed at least 1 post-baseline disease assessment.
Measure: Number; unit: Participants
Groups:
- 2 mg/kg (CLL): CLL patients in MEDI-551 2 mg/kg cohort
- 4 mg/kg (CLL): CLL patients in MEDI-551 4 mg/kg cohort
- 8 mg/kg (CLL): CLL patients in MEDI-551 8 mg/kg cohort
- 12 mg/kg (CLL): CLL patients in MEDI-551 12 mg/kg cohort
Arm/Group | 2 mg/kg (CLL) | 4 mg/kg (CLL) | 8 mg/kg (CLL) | 12 mg/kg (CLL)
Number analyzed (Participants) | 1 | 0 | 0 | 1
Participants | 1 |  |  | 0

16. Secondary Outcome: Number of Participants With Tumour Response in MM Patients
Description: Tumour response is defined as complete response (CR) or partial response (PR) (Durie M et al 2006).
  CR: Negative immunofixation on the serum and urine, and Disappearance of any soft tissue plasmacytomas and 5% or less plasma cells in bone marrow PR: ≥50% reduction of serum M-protein and reduction in 24-h urinary M-protein by ≥90% or to <200mg per 24 h. If the serum and urine M-protein are unmeasurable, a ≥50% decrease in the difference between involved and uninvolved FLC levels is required in place of the M-protein criteria. If serum and urine M-protein are unmeasurable, and serum free light assay is also unmeasurable, ≥50% reduction in plasma cells is required in place of M-protein, provided baseline bone marrow plasma cell percentage was ≥30%. In addition to the above listed criteria, if present at baseline, a ≥50% reduction in the size of soft tissue plasmacytomas is also required.
Time Frame: From the baseline to30 days after the last dose of study drug
Population: All patients with MM who received at least 1 dose of MEDI-551 and completed at least 1 post-baseline disease assessment.
Measure: Number; unit: Participants
Groups:
- 2 mg/kg (MM): MM patients in MEDI-551 2 mg/kg cohort
- 4 mg/kg (MM): MM patients in MEDI-551 4 mg/kg cohort
- 8 mg/kg (MM): MM patients in MEDI-551 8 mg/kg cohort
- 12 mg/kg (MM): MM patients in MEDI-551 12 mg/kg cohort
Arm/Group | 2 mg/kg (MM) | 4 mg/kg (MM) | 8 mg/kg (MM) | 12 mg/kg (MM)
Number analyzed (Participants) | 0 | 1 | 0 | 0
Participants |  | 0 |  |

ADVERSE EVENTS:
Time Frame: AEs were collected throughout the study, from informed consent until the end of 30 days after study treatment. The follow-up period is defined as 3 months after study treatment is discontinued.
Arm/Group | 2 mg/kg | 4 mg/kg | 8 mg/kg | 12 mg/kg
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/7 | 0/4 | 0/6
Other Adverse Events (participants affected / at risk) | 3/3 | 6/7 | 4/4 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 2 mg/kg (N=3) | 4 mg/kg (N=7) | 8 mg/kg (N=4) | 12 mg/kg (N=6)
Epiglottitis (Infections and infestations) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 2 mg/kg (N=3) | 4 mg/kg (N=7) | 8 mg/kg (N=4) | 12 mg/kg (N=6)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 1 | 3 | 3
White blood cell count decreased (Investigations) | 2 | 2 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 2 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 2 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 1 | 4 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 0 | 0
Influenza like illness (General disorders) | 1 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Monarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 0 | 1
Eyelid oedema (Eye disorders) | 0 | 1 | 0 | 0
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Sebaceous adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 2 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No